CLINICAL TRIAL: NCT04787302
Title: A Phase 1, Open-label Trial to Evaluate Target Occupancy of CVL-231 at Muscarinic Receptors Type 4 in Brain Following Single Oral Doses Using Positron Emission Tomography in Healthy Adult Subjects
Brief Title: PET Trial to Evaluate Target Occupancy of CVL-231 on Brain Receptors Following Oral Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CVL-231-1002
Record Dates: First submitted 2021-02-01; First posted 2021-03-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; PET; Healthy Volunteer
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CVL-231 (Experimental)
  Interventions: Drug: CVL-231

INTERVENTIONS:
Drug: CVL-231 — Cohort 1: 30mg dose of CVL-231
  Other Names: PF-06852231
Drug: CVL-231 — Cohort 2: CVL-231 dose to be decided based on results of Cohort 1 or trial may be concluded
  Other Names: PF-06852231
Drug: CVL-231 — Cohort 3: CVL-231 dose to be decided based on results of Cohorts 1 and/or 2
  Other Names: PF-06852231

SUMMARY:
PET Trial to Evaluate Target Occupancy of CVL-231 at Muscarinic Receptors Type 4 in Brain Following Oral Dosing

DETAILED DESCRIPTION:
CVL-231 is a muscarinic acetylcholine receptor (mAChR) activator that selectively binds to the M4 muscarinic receptor subtype (M4 mAChR). CVL-231 is being developed for treatment of psychosis in schizophrenia. The aim of this trial is to characterize the relationship between the M4 receptor occupancy in different regions of the brain following a single oral doses of CVL-231 in healthy adult subjects by positron emission tomography (PET) using the radioligand [11C]MK-6884.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and female subjects of nonchildbearing potential, ages 18 to 55 years, inclusive, at the time of signing the ICF
* Sexually active men with a pregnant or a nonpregnant partner of childbearing potential must agree to use a double-barrier method of birth control, including a condom, and practice contraception during treatment and through 7 days post dose
* Capable of providing informed consent and following study requirements

Exclusion Criteria:

* Subjects who answer yes on the C-SSRS or, in the opinion of the investigator, present a serious risk of suicide
* Subjects with a current history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, hematological, immunological, or neurological disease
* Subjects with a 12-lead ECG demonstrating either of the following (average of 3 ECGs obtained at the Screening Visit):

  * QT interval corrected for heart rate using Fridericia's formula >450 msec
  * Left ventricular hypertrophy
* Orthostatic hypotension, which is defined as a decrease of ≥20 mmHg in systolic blood pressure and/or a decrease of ≥10 mmHg in diastolic blood pressure after at least 3 minutes of standing compared with the immediately previous supine/semi-recumbent blood pressure at Screening or at the prescan time point prior to baseline PET scan.
* Subjects with a current or past personal history of any psychiatric disorder as classified by DSM-5 criteria or immediate family members with any psychiatric disorder as classified by DSM-5 criteria that require treatment
* Subjects with a history of substance or alcohol-use disorder (DSM-5 criteria) within 2 years prior to signing the ICF
* Subjects with other abnormal laboratory test results, vital sign results, or ECG findings
* Subjects who currently use or have used tobacco or nicotine-containing products within 30 days prior to signing the ICF
* Subjects with history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure (5 rem per year)
* Subjects with any anatomical abnormality in the head that would either preclude or tend to confound the analysis of study data, including any clinically significant abnormal findings from MRI of the head
* Current, past or anticipated exposure to radiation in the workplace
* Any subject with a significant acute illness within 7 days prior to administration of study drug or have had a major illness or hospitalization within 1 month prior to administration of study drug
* Any subject who, in the opinion of the sponsor, investigator, or medical monitor, should not participate in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
M4 receptor occupancy in the striatum following single oral doses of CVL-231 in healthy adult subjects | Day 1
  Fraction of M4 receptors occupied by CVL-231 doses

SECONDARY OUTCOMES:
Treatment-emergent adverse events | Upto 9 weeks
Number of subjects with Clinically significant changes in Electrocardiogram | Screening, Pre-scan, Day-1, Day 1 (T=0hour), Day 1 (T=0.5hour), Day 1 (T=3.0hour), Day 2 (T=24hour), Day 10
Number of subjects with clinical significant Clinical laboratory assessments | Screening, Pre-scan, Day-1, Day 2 (T=24hour)
Number of subjects with Clinically significant changes in Vital signs | Screening, Day-1 (T=1hour), Day-1 (T=1.5hour), Day-1, Day 1 (T=0hour), Day 1(T=1.5hour), Day 1 (T=3hour), Day 1 (T=6hr), Day 1 (T=8.0), Day 2 (T-=24hr), Day 10
Number of subjects with clinically significant Physical and neurological examination results | Screening, Day-1 pre-scan, Day-1, Day 2
Suicidality assessed using the Columbia-Suicide Severity Rating Scale | Screening, Day-1, Day 2, Day 10
  Suicidality will be monitored during the trial using the Columbia - Suicide Severity Rating Scale (C-SSRS)
Cmax during scan for CVL-231 | Day 1 (0.5, 1.5 and 2.0 hours)
  Max CVL-231 concentration during PET scan
AUCscan duration for CVL-231 | Day 1 (0.5, 1.5 and 2.0 hours)
  AUC for CVL-231 during PET scan
Cavg/Scan duration for CVL-231 | Day 1 (0.5, 1.5 and 2.0 hours)
  Average CVL-231 concentration during scan
Model estimated Emax and EC50 at M4 receptors in striatum for CVL-231 | Day 1
  Model estimated values for Maximum possible binding (Emax) and CVL-231 concentrations required from hal-maximal binding (EC50)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Leoni, MD, MBA, Study Director — Cerevel Therapeutics, LLC
Locations (2):
- Massachusetts General Hospital Translational and Clinical Research Centers, Boston, Massachusetts, United States
- UZ Leuven, Leuven, Belgium